CLINICAL TRIAL: NCT04551768
Title: An Open-Label Study to Evaluate the Safety and Efficacy of VIRAZOLE® (RIBAVIRIN FOR INHALATION SOLUTION, USP) in Hospitalized Adult Participants With Respiratory Distress Due to COVID-19
Brief Title: Study to Evaluate the Safety and Efficacy of VIRAZOLE® in Hospitalized Adult Participants With Respiratory Distress Due to COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BHC-RIB-5401-GL
Record Dates: First submitted 2020-09-15; First posted 2020-09-16 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 50 mg/mL Virazole (Experimental): 50 mg/mL Virazole aerosolized and administered over 1 hour twice a day for up to 6 days.
  Interventions: Drug: 50 mg/mL Virazole
- 100 mg/mL Virazole (Experimental): 100 mg/mL Virazole aerosolized and administered over 30 minutes twice a day for up to 6 days.
  Interventions: Drug: 100 mg/mL Virazole

INTERVENTIONS:
Drug: 50 mg/mL Virazole — 50 mg/mL Virazole aerosolized and administered over 1 hour twice a day for up to 6 days.
  Arms: 50 mg/mL Virazole
Drug: 100 mg/mL Virazole — 100 mg/mL Virazole aerosolized and administered over 30 minutes twice a day for up to 6 days.
  Arms: 100 mg/mL Virazole

SUMMARY:
This study is a Phase 1, open label, non-randomized, two-arm interventional clinical trial to evaluate the safety and efficacy of Virazole® in hospitalized adult patients who have tested positive for COVID-19 and, as a result, have significant respiratory distress (PaO2/FiO2 ratio <300 mmHg).

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female ≥ 18 years of age.
2. Willing and able to provide written informed consent (or provided by a proxy).
3. Currently hospitalized with laboratory confirmed COVID-19 novel coronavirus infection.
4. PaO2/FiO2 ratio <300 mmHg.
5. Illness of any duration, and at least one of the following:

   * Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), OR
   * Clinical assessment (evidence of rales/crackles on exam) AND SpO2 ≤94% on room air, OR
   * Requiring mechanical ventilation and/or supplemental oxygen.
6. Once released from the hospital, women of childbearing potential (WOCBP) and all men must agree to use at contraception methods for 9 months.

Exclusion Criteria:

1. Pregnant or breast feeding.
2. Respiratory distress for reasons other than COVID-19 infection (e.g., congestive heart failure (CHF), bacterial pneumonia, etc.).
3. Presence of secondary bacterial pneumonia.
4. Presence of significant pulmonary fibrosis.
5. Hypotension (need for hemodynamic pressors to maintain blood pressure).
6. Greater than 7 days on mechanical ventilation.
7. Anemia defined as hemoglobin or RBC <75% of the institutional lower limit of normal for race, age and gender.
8. History of COPD or bronchospasm prior to COVID-19 infection.
9. History of hypersensitivity to ribavirin.
10. Any condition that could cause noncompliance with treatment or may otherwise contraindicate the subject's participation in the study
11. Subject is currently participating in any drug or device clinical investigation.
12. Subject has received an investigational agent or approved drug that, in the Investigator's judgement, may have a chemical or pharmacological interaction with Virazole if administered within 5 half-lives or 30 days of the Baseline Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Change in the clinical status severity (CSS) rating from the first dose date up to the completion of treatment | 7 days
  The severity rating will be based on the ordinal scale of clinical status as follows:
  1. Death.
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices.
  4. Hospitalized, requiring supplemental oxygen.
  5. Hospitalized, not requiring supplemental oxygen.
  6. Not hospitalized, limitation on activities.
  7. Not hospitalized, no limitations on activities.

SECONDARY OUTCOMES:
Time to recover gas exchange to a PaO2/FiO2 ≥300 for at least 24 hours. | 7 days
Time to reach peripheral capillary oxygen saturation (Sp02) >94% for at least 24 hours. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health
Locations (4):
- Greece (3):
  - Bausch Health Site 201, Athens, Attica
  - Bausch Health Site 203, Athens, Attica
  - Bausch Health Site 204, Alexandroupoli, Evros
- Bausch Site 304, Tijuana, Zona Rio, Mexico

IPD SHARING:
Plan to Share IPD: Undecided